



Sponsor's/protocol number: 20HH5790

NCT number:

| IR | IRAS Project ID: 277754 | |
|---|---|---|
| | CONSENT FORM | -<br>- |
| Ti | tle of Project: The evaluation of the pathophysiology of Varicose veins in pregnancy | |
| Na | ame of Researcher: Dr. M. Aslam | |
| | Please initial all boxe | s |
| 1. | I confirm that I have read and understand the subject information sheet dated <b>16 May 2021</b> version <b>2</b> for the above study and have had the opportunity to ask questions which have been answered fully. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without medical care or legal rights being affected. | |
| 3. | I understand that relevant sections of medical notes and data collected during the study may be looked at by individuals from the Sponsor, the NHS and the research team, including regulatory authorities, monitors and auditors, where it is relevant to my participation in this research. I give permission for these individuals to have access to these records. | |
| 4. | I agree to my GP being informed of my participation in the study. | |
| 5. | I understand that all information will remain confidential. | |
| 6. | I voluntarily give consent to participate in this study. | |
| 7. | I give/ do not give consent for information collected about me to be used to support other research in the future, including those outside of the EEA. | |
| | ☐ Yes ☐ No | |

## Imperial College Healthcare NHS Trust Imperial College London

| I give/ do not give consent for samples collected during this study to be used in future ethically approved studies. | | | |
|---|---|---|---|
| Yes | | No | |
| <ol><li>I give/ do not give permission for<br/>including these outsides of the E</li></ol> | | other organisations, | |
| Yes | | No | |
| <b>10</b> . I give consent for my blood samր | oles in this study to be use | d for genetic testing. | |
| <b>11.</b> I agree that any significant incid withdrawn from the study. | ental findings will be refer | red to my clinician and I will b | е |
| <b>12.</b> I agree to receive a lay summar study finishes by email or letter. | y of the research study res | sults after the research | |
| Yes | | No | |
| <b>13.</b> I give consent to being contacte studies. | d to potentially taking part | in other research | |
| Yes | | No | |
| Print Name of Participant | <br>Date | Signature | |
| Print Name of Person taking Consent | Date | Signature | |

When completed, 1 for patient; 1 for researcher site file; 1 (original) to be kept in medical notes

IRAS ID: **277754** V2.0 16 May 2021 © Imperial College of Science, Technology and Medicine